CLINICAL TRIAL: NCT03502122
Title: Design and Verification of Individualized Smart Assistive Devices for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Central University, Taiwan (Other)
Responsible Party: Principal Investigator, Chun-Chuan Chen, Associate professor, National Central University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201012009IA
Record Dates: First submitted 2018-03-31; First posted 2018-04-18 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Stroke
Keywords: stroke; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR rehabilitation (Experimental): Virtual Reality based rehabilitation therapy for motor function, 1 hour a time at an intensity of three times per week over 8 weeks (total, 24 sessions).
  Interventions: Other: VR rehabilitation for motor function
- control- conventional rehabilitation (Active Comparator): conventional rehabilitation therapy for motor function, 1 hour a time at an intensity of three times per week over 8 weeks (total, 24 sessions).
  Interventions: Other: VR rehabilitation for motor function

INTERVENTIONS:
Other: VR rehabilitation for motor function — rehabilitation for motor function
  Other Names: VR rehabilitation therapy

SUMMARY:
This study aims to design and verify a multi-mode smart assistive device system for Stroke Rehabilitation by using EEG, fMRI, IMU and questioners

ELIGIBILITY:
Inclusion Criteria:

* the first time hemiparetic stroke;
* diagnosis confirmed by a physician on the basis of the findings of neurological examinations and brain imaging (magnetic resonance imaging or computed tomography scan);
* aged between 20 and 85 years;
* Brunnstrom's stage II to V over the proximal and distal part of the upper extremity on the affected side;
* no cognitive dysfunction, measured by the Mini-Mental State Exam (≧24; suggested by 36 with respect to age and educational level)
* willing/able to participate and having signed an informed consent form.

Exclusion Criteria:

* unstable vital sign
* irreversible contracture over any of the joints of the affected upper extremity
* history of surgery, fracture, arthritis, pain, or any other complications that might influence the recovery of upper extremity function like aphasia, apraxia and neglect;
* having spasticity, as measured using the Modified Ashworth scale (score > 2);
* poststroke seizure;
* heart attack within 3 months poststroke; cortical lesions in any of the five core motor areas of interest, including the bilateral M1, the bilateral PM, and the SMA.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04-24 (Actual); Primary Completion 2014-05-28 (Actual); Study Completion 2014-05-28 (Actual)

PRIMARY OUTCOMES:
Change in FUGL- MEYER ASSESSMENT OF PHYSICAL PERFORMANCE (FMA) | pre, post (after 24 hrs of intervention) and follow-up (one month after finishing intervention )
  FUGL- MEYER ASSESSMENT OF PHYSICAL PERFORMANCE (FMA)

SECONDARY OUTCOMES:
change in upper extremity performance evaluation test for the elderly (TEMPA) | pre, post (after 24 hrs of intervention) and follow-up (one month after finishing intervention )
  upper extremity performance evaluation test for the elderly (TEMPA)
change in Brunnstrom stage | pre, post (after 24 hrs of intervention) and follow-up (one month after finishing intervention )
  Brunnstrom stage
change in Wolf motor function | pre, post (after 24 hrs of intervention) and follow-up (one month after finishing intervention )
  Wolf motor function

IPD SHARING:
Plan to Share IPD: Undecided
undecided .